CLINICAL TRIAL: NCT01713894
Title: Utility of a Clinically Relevant Decision Aid, for Parents Facing Extremely Premature Delivery
Brief Title: Decision Aid - Extreme Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Virtua Health (Other); University of Michigan (Other); Endeavor Health (Other)
Responsible Party: Principal Investigator, Ursula Guillen, Principal Investigator; Assistant Professor, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Decision Aid - Prematurity
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Prematurity; Decision Support
Keywords: Counseling; Limits of viability
MeSH Terms: conditions — Premature Birth | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Other): In this arm of the study, parents will be counseled using a decision aid.
  Interventions: Other: Decision Aid
- Standard (Other): In this arm of the study, parents will be counseled using current standard methods.
  Interventions: Other: Standard

INTERVENTIONS:
Other: Decision Aid
  Arms: Decision Aid
Other: Standard
  Arms: Standard

SUMMARY:
The purpose of this study is to assess in a pilot randomized controlled trial the following PICOT question: In parents facing extreme premature delivery, does the use of an existing validated visual decision aid as compared to standard counseling, reduce the primary outcome of parental decisional conflict? Furthermore, is such a decision aid understood and applicable across differing populations of different ethnic backgrounds and social classes?

ELIGIBILITY:
Inclusion Criteria:

* physicians who counsel women at the limits of viability
* women who are receiving counseling at the limits of viability

Exclusion Criteria:

* Known congenital malformations or lethal anomalies, still birth in which the fetuses' death was known before labor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05; Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | within 1 week after consult
  Decisional conflict is the state of uncertainty about the course of action to take when making choices involving risk or uncertainty of outcomes. Decisional conflict is assessed using the Decisional Conflict Scale

SECONDARY OUTCOMES:
Knowledge | within 1 week after consult

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Guillen, MD, Principal Investigator — Christiana Care Health Systems
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

REFERENCES:
- [Derived] Guillen U, Mackley A, Laventhal N, Kukora S, Christ L, Derrick M, Batza J, Ghavam S, Kirpalani H. Evaluating the Use of a Decision Aid for Parents Facing Extremely Premature Delivery: A Randomized Trial. J Pediatr. 2019 Jun;209:52-60.e1. doi: 10.1016/j.jpeds.2019.02.023. Epub 2019 Apr 2. PMID 30952510